CLINICAL TRIAL: NCT02418208
Title: Clinical Trial Protocol for the Establishment of Normative Data of Brain Network Activation (BNA) Using Evoked Response Potentials in Adolescents, Young Adults and Adults
Brief Title: Normative Data Base of Brain Network Activation (BNA) Using Evoked Response Potentials
Acronym: Normative
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-25
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Normative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test retest- 2 visits: Eligible participants will arrive for 2 testing visits a week apart and an optional third visit within 6-12 months.
  Interventions: Diagnostic Test: Performint EEG tests and BNA analysis
- Single Visit: Eligible participants will arrive for a single testing visit
  Interventions: Diagnostic Test: Performint EEG tests and BNA analysis

INTERVENTIONS:
Diagnostic Test: Performint EEG tests and BNA analysis

SUMMARY:
Purpose: EEstablish normative data of ElMindA's Brain Network Activation (BNA) using evoked response potentials in adolescents, young adults and Adults.

Trial design: Open, one-arm, prospective, age-stratified, multi site. Enrollment size: Up to 1500 subjects will be enrolled in 4 or more sites. Study duration: Each patient will be followed up for up to 1 year. Overall study duration will be up to 1.5 years. Patient population: Adolescents, young adults and Adults of both genders.

Age range:

* 10-11.99
* 12-13.99
* 14-15.99
* 16-17.99
* 18-24.99
* 25-29.99
* 30-34.99
* 35-39.99
* 40-44.99
* 45-49.99
* 50-54.99
* 55-60
* 60 and above

Objective: Establishment of normative data of BNA.

DETAILED DESCRIPTION:
Currently, there is no reliable, bedside, and non-invasive method for assessing connectivity changes in electrophysiological activity of the brain associated with brain-related pathologies, e.g., concussion, ADHD, autistic spectrum disorders (ASD), etc. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a non-invasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA) to temporally and spatially map brain function, connectivity and synchronization.

The need of objective measures that will help the clinician in its decision making in brain-related pathologies is recognized. BNA is a new imaging modality that has been developed to fill this gap.

ELIGIBILITY:
Inclusion criteria:

1. Age 10-years and above.
2. Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments.
3. Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self).

Exclusion criteria:

1. Has participated in the past 6 months in an organized contact sport activity (e.g., football, hockey, soccer, rugby, lacrosse, martial arts, Boxing).
2. Currently with lice or open wounds on scalp.
3. Any chronic disease or condition which affects the nervous system as determined by clinical neurological evaluation, medical history or PI discretion.
4. Active (within 1 month) Migraine history or clinically significant reoccurring Migraine episodes.
5. Any psychiatric disorder, e.g., depression, bipolar disorder, schizophrenic disorder, etc. as determined by clinical evaluation and the Mini International Neuropsychiatric Interview (MINI)
6. Any CNS neurologic disorder, e.g., epilepsy, seizures, etc. as determined by clinical evaluation
7. Any neuropsychological disorders, e.g.: ADHD, Autistic Spectrum Disorder (ASD), etc. as determined by clinical evaluation
8. History of Special education, e.g., reading disorder (dyslexia), writing disorder (dysgraphia), math disorder (dyscalculia), nonverbal learning disorder.
9. History of any medication affecting CNS within the last 3 months, e.g., antidepressants, anticonvulsants, psychostimulants, first generation antihistamines, etc. The investigator should consider including subjects which had used such drugs for a short period according to a logical calculation of the drug's half-life.
10. Substance abuse in the last 3 months and any clinically significant substance dependency as determined by the MINI evaluation and PI discretion.
11. Significant sensory deficits, e.g., deafness or blindness.
12. Pregnant women or women that are 1 month following a childbirth.
13. History of any clinically significant brain trauma as determined by the investigator.
14. History of more than 1 clinically diagnosed concussion.
15. Clinically diagnosed with a concussion in the past year. Minor deviations to eligibility criteria may be made on a case-by-case basis prior to enrollment if approved by the Sponsor, in writing, in agreement with the Investigator.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 1500 subjects, from both genders, aged 10 years and above will be recruited, stratified to age groups.
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Developing a BNA database for normative population. | 1.5 years
  Functional networks of brain activity in healthy individuals measured using analysis of EEG Event Related Potential (ERP) data

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Clinical trials of the Rockies, Inc., Denver, Colorado
  - Psychiatric Medicine Associates, Llc, Skokie, Illinois
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Ohio Clinical Trials, Inc., Columbus, Ohio
- Cytespace Research Private Limited, Banglore, India